CLINICAL TRIAL: NCT03214588
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm Study to Evaluate Efficacy, Tolerability, and Pharmacokinetics of Multiple Doses of Oral TAK-831 in Adult Subjects With Friedreich Ataxia
Brief Title: Efficacy, Tolerability, and Pharmacokinetics of Multiple Doses of Oral TAK-831 in Adults With Friedreich Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-831-1501; U1111-1189-7951 (Registry Identifier: WHO)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Friedreich Ataxia
Keywords: Drug Therapy
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): TAK-831 placebo-matching tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: TAK-831 Placebo
- TAK-831 75 mg (Experimental): TAK-831 75 mg, tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: TAK-831
- TAK-831 300 mg (Experimental): TAK-831 300 mg, tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: TAK-831

INTERVENTIONS:
Drug: TAK-831 — TAK-831 tablets
  Arms: TAK-831 300 mg; TAK-831 75 mg
Drug: TAK-831 Placebo — TAK-831 placebo matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK-831 versus placebo on upper extremity (arm and hands) motor function and manual dexterity. This study will also evaluate the efficacy of TAK-831 versus placebo on activities of daily living (ADL) and other secondary assessments.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. TAK-831 is being tested to treat people who have Friedreich ataxia. This study will look at upper extremity (arms and hands) motor function and manual dexterity of people who take TAK-831. Efficacy evaluations also include other neurological, functional, and patient performance assessments.

The study will enroll approximately 65 participants. Participants will be randomly assigned in a 2:1:2 ratio to one of the three treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-831 High dose
* TAK-831 Low dose
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will be asked to take three tablets of high dose, low dose, or placebo twice a day for 12 weeks.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 13 weeks. Participants will make 5 visits to the clinic, and will be contacted by telephone for an exit interview no later than 7 days after their final visit or termination. Participants will also receive a safety follow-up phone call 7 to 17 days after receiving their last dose of TAK-831.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a genetically-confirmed diagnosis (homozygous for guanine-adenine-adenine [GAA] repeat expansions in the frataxin gene [FXN] in the affected range of Friedreich ataxia [FRDA] or a compound heterozygous expansion with a point mutation or deletion), with an established disease stage of 2 to 5, inclusive, as determined by the Functional Staging for Ataxia, at Screening.

Key Exclusion Criteria:

1. Received a diagnosis of ataxic syndromes other than FRDA.
2. Has a history of cancer, except basal cell carcinoma or in situ cervical cancer that has been in remission for greater than or equal to (>=5) years prior to first dose of study drug.
3. Known to be currently infected or has been infected with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
4. Has a known hypersensitivity to any component of the formulation of TAK-831.
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse.
6. Has taken any excluded medication, or has had insufficient washout of medications or is unable or unwilling to discontinue medications as required by the protocol.
7. If male, the participant intends to donate sperm during the course of this study or for 95 days after the last dose of study drug.
8. If female, the participant is of childbearing potential and lactating, pregnant (positive prerandomization serum pregnancy test), or plans to become pregnant before participating in the study, during the study, or within 35 days after last dose of the study drug, or intending to donate ova during such time period.
9. Has a history of neuroleptic malignant syndrome, water intoxication, or paralytic ileus or other conditions that may interfere with absorption of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Ataxia Center, Los Angeles, California
  - University of Florida Center for Movement Disorders, Gainesville, Florida
  - USF College of Medicine, Tampa, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 08 November 2017 to 27 December 2018.
Pre-assignment Details: Participants with a diagnosis of Friedreich Ataxia were randomized in a 2:1:2 ratio to receive TAK-831 75 mg TAK-831 300 mg or TAK-831 placebo-matching tablets twice daily.
Period: Overall Study
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Started | 27 | 14 | 26
Completed | 26 | 13 | 24
Not Completed | 1 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Reason Not Specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study drug for the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg | Total
Number analyzed (Participants) | 27 | 14 | 26 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (11.01) | 31.1 (11.28) | 29.6 (8.92) | 31.1 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 15 | 37
  Male | 10 | 9 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 27 | 13 | 26 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight(kg)/[height(m)^2]
  kg/m^2 | 24.89 (4.920) | 24.94 (4.400) | 23.02 (3.862) | 24.18 (4.456)
Average Inverse Time to Complete 9-hole peg test (9-HPT-1) [Median (Full Range); unit: 1/seconds] — The inverse of the time to complete the 9-hole peg test (9-HPT-1), defined as 1/(time to complete the 9-hole peg test), is summarized.
  1/seconds
    First Assessment | 0.01740 [0.0055 to 0.0298] | 0.01660 [0.0062 to 0.0278] | 0.01575 [0.0075 to 0.0404] | 0.01680 [0.0055 to 0.0404]
    Second Assessment | 0.01710 [0.0082 to 0.0254] | 0.01605 [0.0073 to 0.0269] | 0.01595 [0.0067 to 0.0391] | 0.01660 [0.0067 to 0.0391]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Inverse Time to Complete the 9-Hole Peg Test (9-HPT-1)
Description: The 9-HPT-1 is a measure of timed upper extremity (arm and hand) function and manual dexterity. The participant picks up pegs 1 at a time (9 in total), using 1 hand only, and places them into holes on the board as quickly as possible, in any order until all holes are filled. Then, without pausing, the participant removes the pegs 1 at a time and returns them as quickly as possible. Each participant performs this task twice with each hand separately. Results on both tests are then averaged for an overall task completion time and the inverse transform is performed. A positive change from Baseline indicates improvement. Change from Baseline in 9-HPT-1 was analyzed using mixed model for repeated measures (MMRM) analysis of covariance (ANCOVA) with Baseline 9-HPT-1 as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline 9-HPT-1-by-visit interactions.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) included all randomized participant who received at least 1 dose of the study drug for the treatment period. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: 1/seconds
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 24 | 12 | 24
1/seconds | 0.00038 (0.000448) | -0.00017 (0.000622) | -0.00032 (0.000445)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p > 0.999, ANCOVA — P-values are 1-sided, with the alternative hypothesis that TAK-831 is superior to placebo in the clinically favorable direction; Least Squares Mean Difference = -0.00054, 90% CI 2-sided [-0.00179 to 0.00070], Standard Error of Mean 0.000746
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p > 0.999, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.00069, 90% CI 2-sided [-0.00172 to 0.00033], Standard Error of Mean 0.000616

2. Secondary Outcome: Change From Baseline in the Activities of Daily Living (ADL) Component Score of the Friedreich Ataxia Rating Scale (FARS)
Description: The ADL component of the FARS includes 9 subscales: speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function. Each of these subscales is rated on a 5-point scale where 0=normal to 4=severe disability/inability to carry out activity independently for a total possible score of 0 to 36, with higher scores representing greater disability/dependency. A negative change from Baseline indicates improvement. Change from Baseline in FARS ADL upper limb function items were analyzed using MMRM ANCOVA with Baseline FARS ADL as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline FARS ADL-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7 and 12
Population: FAS included all randomized participant who received at least 1 dose of the study drug for the treatment period. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 27 | 13 | 26
  Change from Baseline at Week 2 | -0.25 (0.468) | -1.12 (0.665) | 0.34 (0.463)
  Change from Baseline at Week 7: number analyzed (Participants) | 26 | 13 | 24
  Change from Baseline at Week 7 | -0.33 (0.465) | -0.15 (0.655) | 0.03 (0.467)
  Change from Baseline at Week 12: number analyzed (Participants) | 24 | 12 | 24
  Change from Baseline at Week 12 | -0.61 (0.493) | -0.37 (0.696) | -0.24 (0.488)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.135, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.87, 90% CI 2-sided [-2.18 to 0.44], Standard Error of Mean 0.782
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.818, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.59, 90% CI 2-sided [-0.48 to 1.66], Standard Error of Mean 0.640
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.591, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.18, 90% CI 2-sided [-1.11 to 1.47], Standard Error of Mean 0.770
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.713, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.36, 90% CI 2-sided [-0.71 to 1.44], Standard Error of Mean 0.643
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.616, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.24, 90% CI 2-sided [-1.13 to 1.62], Standard Error of Mean 0.822
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.708, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.37, 90% CI 2-sided [-0.76 to 1.51], Standard Error of Mean 0.679

3. Secondary Outcome: Change From Baseline in the Inverse Time to Complete the 9-HPT-1
Description: The 9-HPT-1 is a measure of timed upper extremity (arm and hand) function and manual dexterity. The participant picks up pegs 1 at a time (9 in total), using 1 hand only, and places them into holes on the board as quickly as possible, in any order until all holes are filled. Then, without pausing, the participant removes the pegs 1 at a time and returns them as quickly as possible. Each participant performs this task twice with each hand separately. Results on both tests are then averaged for an overall task completion time, and the inverse transform is performed. A positive change from Baseline indicates improvement. Change from Baseline in 9-HPT-1 was analyzed using MMRM ANCOVA with Baseline 9-HPT-1 as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline 9-HPT-1-by-visit interactions.
Time Frame: Baseline and Weeks 2 and 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: 1/seconds
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
1/seconds
  Change from Baseline at Week 2 | 0.00087 (0.000371) | 0.00048 (0.000508) | -0.00006 (0.000370)
  Change from Baseline at Week 7: number analyzed (Participants) | 26 | 13 | 24
  Change from Baseline at Week 7 | 0.00040 (0.000462) | 0.00026 (0.000643) | -0.00004 (0.000471)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.741, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.00039, 90% CI 2-sided [-0.00140 to 0.00062], Standard Error of Mean 0.000604
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.964, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.00093, 90% CI 2-sided [-0.00177 to -0.00008], Standard Error of Mean 0.000505
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.573, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.00014, 90% CI 2-sided [-0.00143 to 0.00115], Standard Error of Mean 0.000772
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.749, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.00044, 90% CI 2-sided [-0.00152 to 0.00064], Standard Error of Mean 0.000646

4. Secondary Outcome: Change From Baseline in the ADL Component Individual Item Scores
Description: The ADL component of the FARS includes 9 subscales: speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function. Each of these subscales is rated on a 5-point scale where 0=normal to 4=severe disability/inability to carry out activity independently. A negative change from Baseline indicates improvement. Statistical analyses were available for the following subscales: cutting food-handling utensils, dressing and personal hygiene.
Time Frame: Baseline and Weeks 2, 7 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change at Week 2, Speech: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Speech | 0.07 (0.494) | -0.15 (0.427) | -0.06 (0.432)
  Change at Week 7, Speech: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Speech | 0.06 (0.516) | -0.08 (0.400) | -0.15 (0.429)
  Change at Week 12, Speech: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Speech | 0.06 (0.425) | -0.17 (0.492) | -0.02 (0.403)
  Change at Week 2, Swallowing: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Swallowing | 0.00 (0.555) | 0.04 (0.320) | -0.19 (0.618)
  Change at Week 7, Swallowing: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Swallowing | 0.04 (0.422) | 0.08 (0.534) | -0.06 (0.756)
  Change at Week 12, Swallowing: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Swallowing | -0.15 (0.403) | 0.13 (0.311) | -0.27 (0.589)
  Change at Week 2, Cutting-Handling Utensils: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Cutting-Handling Utensils | -0.13 (0.451) | -0.04 (0.380) | 0.12 (0.535)
  Change at Week 7, Cutting-Handling Utensils: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Cutting-Handling Utensils | -0.21 (0.619) | -0.15 (0.240) | 0.08 (0.525)
  Change at Week 12, Cutting-Handling Utensils: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Cutting-Handling Utensils | -0.19 (0.548) | -0.08 (0.417) | 0.08 (0.482)
  Change at Week 2, Dressing: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Dressing | 0.00 (0.392) | -0.12 (0.506) | 0.12 (0.516)
  Change at Week 7, Dressing: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Dressing | 0.04 (0.372) | 0.04 (0.380) | -0.04 (0.292)
  Change at Week 12, Dressing: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Dressing | 0.02 (0.561) | -0.04 (0.498) | -0.10 (0.361)
  Change at Week 2, Personal Hygiene: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Personal Hygiene | -0.02 (0.427) | 0.00 (0.456) | 0.15 (0.485)
  Change at Week 7, Personal Hygiene: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Personal Hygiene | 0.08 (0.659) | 0.19 (0.560) | 0.04 (0.530)
  Change at Week 12, Personal Hygiene: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Personal Hygiene | 0.08 (0.602) | 0.21 (0.656) | 0.06 (0.517)
  Change at Week 2, Falling: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Falling | 0.06 (0.560) | 0.04 (0.660) | 0.02 (0.435)
  Change at Week 7, Falling: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Falling | -0.13 (0.481) | 0.54 (1.266) | -0.04 (0.706)
  Change at Week 12, Falling: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Falling | -0.29 (0.932) | 0.50 (0.739) | -0.33 (0.856)
  Change at Week 2, Walking: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Walking | -0.02 (0.470) | -0.08 (0.494) | 0.08 (0.272)
  Change at Week 7, Walking: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Walking | 0.00 (0.245) | -0.08 (0.344) | -0.06 (0.450)
  Change at Week 12, Walking: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Walking | 0.13 (0.516) | -0.08 (0.557) | 0.02 (0.179)
  Change at Week 2, Quality of Sitting Position: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Quality of Sitting Position | 0.09 (0.605) | -0.31 (0.663) | 0.10 (0.375)
  Change at Week 7, Quality of Sitting Position: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Quality of Sitting Position | 0.06 (0.497) | -0.27 (0.753) | 0.00 (0.511)
  Change at Week 12,Quality of Sitting Position: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12,Quality of Sitting Position | 0.10 (0.589) | -0.33 (0.778) | 0.08 (0.458)
  Change at Week 2, Bladder Function: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Bladder Function | -0.09 (0.555) | -0.27 (0.439) | 0.13 (0.460)
  Change at Week 7, Bladder Function: number analyzed (Participants) | 26 | 13 | 24
  Change at Week 7, Bladder Function | -0.08 (0.643) | -0.15 (0.555) | 0.08 (0.381)
  Change at Week 12, Bladder Function: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Bladder Function | -0.17 (0.504) | -0.42 (0.557) | -0.04 (0.550)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Cutting-Handling Utensils; Test type: Superiority; p = 0.571, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.03, 90% CI 2-sided [-0.23 to 0.29], Standard Error of Mean 0.154 — MMRM ANCOVA with Baseline FARS ADL as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline FARS ADL-by-visit interactions
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Cutting-Handling Utensils; Test type: Superiority; p = 0.963, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.23, 90% CI 2-sided [0.02 to 0.44], Standard Error of Mean 0.126 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Cutting-Handling Utensils; Test type: Superiority; p = 0.515, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.01, 90% CI 2-sided [-0.27 to 0.28], Standard Error of Mean 0.165 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Cutting-Handling Utensils; Test type: Superiority; p = 0.986, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.31, 90% CI 2-sided [0.08 to 0.54], Standard Error of Mean 0.138 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Cutting-Handling Utensils; Test type: Superiority; p = 0.718, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.09, 90% CI 2-sided [-0.18 to 0.37], Standard Error of Mean 0.162 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Cutting-Handling Utensils; Test type: Superiority; p = 0.986, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.30, 90% CI 2-sided [0.08 to 0.52], Standard Error of Mean 0.133 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Dressing; Test type: Superiority; p = 0.153, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.15, 90% CI 2-sided [-0.40 to 0.09], Standard Error of Mean 0.148 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Dressing; Test type: Superiority; p = 0.861, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.13, 90% CI 2-sided [-0.07 to 0.33], Standard Error of Mean 0.119 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Dressing; Test type: Superiority; p = 0.443, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.02, 90% CI 2-sided [-0.22 to 0.18], Standard Error of Mean 0.120 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Dressing; Test type: Superiority; p = 0.359, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.04, 90% CI 2-sided [-0.20 to 0.13], Standard Error of Mean 0.100 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Dressing; Test type: Superiority; p = 0.268, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.10, 90% CI 2-sided [-0.36 to 0.17], Standard Error of Mean 0.157 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Dressing; Test type: Superiority; p = 0.411, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.03, 90% CI 2-sided [-0.24 to 0.19], Standard Error of Mean 0.129 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Personal Hygiene; Test type: Superiority; p = 0.358, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.06, 90% CI 2-sided [-0.31 to 0.20], Standard Error of Mean 0.151 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Personal Hygiene; Test type: Superiority; p = 0.946, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.20, 90% CI 2-sided [0.00 to 0.41], Standard Error of Mean 0.123 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Personal Hygiene; Test type: Superiority; p = 0.505, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.32 to 0.33], Standard Error of Mean 0.193 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Personal Hygiene; Test type: Superiority; p = 0.658, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.06, 90% CI 2-sided [-0.20 to 0.33], Standard Error of Mean 0.158 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Personal Hygiene; Test type: Superiority; p = 0.649, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.24 to 0.38], Standard Error of Mean 0.184 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Personal Hygiene; Test type: Superiority; p = 0.661, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.06, 90% CI 2-sided [-0.19 to 0.32], Standard Error of Mean 0.151 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in the Modified Friedreich Ataxia Rating Scale Neurological Examination (mFARS-neuro) Total Score
Description: The mFARS-neuro neurological examination is a clinician-rated measure based on neural substrates affected in Friedreich ataxia including: bulbar on a scale of 0-11, upper limb coordination on a scale of 0-36, lower limb coordination on a scale of 0-16, and upright stability/gait functions on a scale of 0-36 for a total possible score of 0 to 99 with higher scores representing greater disability. A negative change from Baseline indicates improvement. Change from Baseline in mFARS-neuro was analyzed using MMRM ANCOVA with Baseline mFARS-neuro as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline mFARS-neuro-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 27 | 13 | 26
  Change from Baseline at Week 2 | -3.36 (0.650) | -0.70 (0.919) | -0.58 (0.647)
  Change from Baseline at Week 7: number analyzed (Participants) | 26 | 13 | 23
  Change from Baseline at Week 7 | -2.41 (0.799) | -2.01 (1.114) | -1.35 (0.828)
  Change from Baseline at Week 12: number analyzed (Participants) | 24 | 12 | 24
  Change from Baseline at Week 12 | -3.30 (0.762) | -1.28 (1.057) | -1.19 (0.752)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.992, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 2.67, 90% CI 2-sided [0.86 to 4.47], Standard Error of Mean 1.078
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.999, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 2.78, 90% CI 2-sided [1.29 to 4.28], Standard Error of Mean 0.892
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.616, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.40, 90% CI 2-sided [-1.84 to 2.64], Standard Error of Mean 1.338
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.823, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 1.06, 90% CI 2-sided [-0.83 to 2.95], Standard Error of Mean 1.131
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.942, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 2.02, 90% CI 2-sided [-0.10 to 4.13], Standard Error of Mean 1.266
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.975, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 2.11, 90% CI 2-sided [0.35 to 3.87], Standard Error of Mean 1.053

6. Secondary Outcome: Change From Baseline in the mFARS-neuro Subscales Scores
Description: The mFARS-neuro neurological examination is a clinician-rated measure based on neural substrates affected in Friedreich ataxia including: bulbar on a scale of 0-11, upper limb coordination on a scale of 0-36, lower limb coordination on a scale of 0-16, and upright stability/gait functions on a scale of 0-36, with the higher scores representing greater disability. A negative change from Baseline indicates improvement. Change from Baseline in mFARS-neuro was analyzed using MMRM ANCOVA with Baseline mFARS-neuro as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline mFARS-neuro-by visit interactions.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
unit on a scale
  Change at Week 2, Bulbar: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Bulbar | 0.08 (0.080) | 0.15 (0.112) | 0.14 (0.082)
  Change at Week 7, Bulbar: number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Bulbar | 0.01 (0.074) | -0.08 (0.102) | 0.17 (0.079)
  Change at Week 12, Bulbar: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Bulbar | 0.01 (0.085) | 0.06 (0.118) | 0.21 (0.087)
  Change at Week 2, Upper Limb Coordination: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Upper Limb Coordination | -1.55 (0.425) | 0.44 (0.601) | -0.53 (0.419)
  Change at Week 7, Upper Limb Coordination: number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Upper Limb Coordination | -0.90 (0.533) | 0.17 (0.741) | -0.72 (0.547)
  Change at Week 12, Upper Limb Coordination: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Upper Limb Coordination | -1.19 (0.608) | 0.02 (0.848) | -0.65 (0.602)
  Change at Week 2, Lower Limb Coordination: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Lower Limb Coordination | -0.92 (0.292) | -0.52 (0.415) | -0.14 (0.289)
  Change at Week 7, Lower Limb Coordination: number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Lower Limb Coordination | -0.84 (0.494) | -0.88 (0.691) | -0.67 (0.516)
  Change at Week 12, Lower Limb Coordination: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Lower Limb Coordination | -1.62 (0.449) | -0.63 (0.625) | -0.67 (0.445)
  Change at Week 2, Upright Stability: number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Upright Stability | -0.5 (0.37) | -0.3 (0.53) | 0.5 (0.38)
  Change at Week 7, Upright Stability: number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Upright Stability | -0.2 (0.27) | -0.8 (0.38) | 0.4 (0.28)
  Change at Week 12, Upright Stability: number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Upright Stability | -0.1 (0.35) | -0.3 (0.48) | 0.4 (0.34)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Bulbar; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.15 to 0.29], Standard Error of Mean 0.133
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Bulbar; Test type: Superiority; Least Squares Mean Difference = 0.06, 90% CI 2-sided [-0.12 to 0.25], Standard Error of Mean 0.110
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Bulbar; Test type: Superiority; Least Squares Mean Difference = -0.10, 90% CI 2-sided [-0.30 to 0.11], Standard Error of Mean 0.122
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Bulbar; Test type: Superiority; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-0.02 to 0.33], Standard Error of Mean 0.104
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Bulbar; Test type: Superiority; Least Squares Mean Difference = 0.05, 90% CI 2-sided [-0.19 to 0.28], Standard Error of Mean 0.141
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Bulbar; Test type: Superiority; Least Squares Mean Difference = 0.20, 90% CI 2-sided [0.00 to 0.40], Standard Error of Mean 0.118
Statistical Analysis 7: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 1.99, 90% CI 2-sided [0.83 to 3.14], Standard Error of Mean 0.689
Statistical Analysis 8: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 1.02, 90% CI 2-sided [0.06 to 1.97], Standard Error of Mean 0.571
Statistical Analysis 9: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 1.08, 90% CI 2-sided [-0.40 to 2.55], Standard Error of Mean 0.882
Statistical Analysis 10: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.18, 90% CI 2-sided [-1.06 to 1.43], Standard Error of Mean 0.743
Statistical Analysis 11: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 1.21, 90% CI 2-sided [-0.48 to 2.91], Standard Error of Mean 1.016
Statistical Analysis 12: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Upper Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.53, 90% CI 2-sided [-0.87 to 1.94], Standard Error of Mean 0.840
Statistical Analysis 13: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.40, 90% CI 2-sided [-0.41 to 1.20], Standard Error of Mean 0.482
Statistical Analysis 14: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.79, 90% CI 2-sided [0.12 to 1.45], Standard Error of Mean 0.397
Statistical Analysis 15: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = -0.04, 90% CI 2-sided [-1.44 to 1.36], Standard Error of Mean 0.837
Statistical Analysis 16: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.17, 90% CI 2-sided [-1.01 to 1.36], Standard Error of Mean 0.707
Statistical Analysis 17: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.99, 90% CI 2-sided [-0.27 to 2.25], Standard Error of Mean 0.755
Statistical Analysis 18: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Lower Limb Coordination; Test type: Superiority; Least Squares Mean Difference = 0.95, 90% CI 2-sided [-0.09 to 2.00], Standard Error of Mean 0.626
Statistical Analysis 19: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Upright Stability; Test type: Superiority; Least Squares Mean Difference = 0.2, 90% CI 2-sided [-0.8 to 1.3], Standard Error of Mean 0.63
Statistical Analysis 20: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Upright Stability; Test type: Superiority; Least Squares Mean Difference = 1.0, 90% CI 2-sided [0.1 to 1.9], Standard Error of Mean 0.52
Statistical Analysis 21: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Upright Stability; Test type: Superiority; Least Squares Mean Difference = -0.5, 90% CI 2-sided [-1.3 to 0.2], Standard Error of Mean 0.45
Statistical Analysis 22: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Upright Stability; Test type: Superiority; Least Squares Mean Difference = 0.6, 90% CI 2-sided [0.0 to 1.2], Standard Error of Mean 0.38
Statistical Analysis 23: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Upright Stability; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-1.2 to 0.7], Standard Error of Mean 0.57
Statistical Analysis 24: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Upright Stability; Test type: Superiority; Least Squares Mean Difference = 0.5, 90% CI 2-sided [-0.3 to 1.3], Standard Error of Mean 0.48

7. Secondary Outcome: Change From Baseline in the mFARS-neuro Individual Item Scores
Description: mFARS-neuro examination is a clinician-rated measure based on neural substrates affected in Friedreich ataxia individual items:Cough,Speech,Right(R)Finger to Finger Test,Left(L)Finger to Finger Test,R-Nose to Finger Test,L-Nose to Finger Test,R-Dysmetria Test,L-Dysmetria Test,Rapid Alternating Movement(RAM)of R-Hands,RAM of L-Hands,R-Finger Taps(FT),L-FT,R-Heel Along Shin Slide,L-Heel Along Shin Slide,R-Heel Along Shin Tap,L-Heel Along Shin Tap,Siting Posture,Stance Feet Apart(SFA)-3 Trial Average(TTA),SFA(Eyes Closed)-TTA,Stance Feet Together(SFT)-TTA,SFT(Eyes Closed)-TTA,Tandem Stance-TTA,Stance on Dominant Foot-TTA,Tandem Walk and Gait.Items were scored on scale of 0 to 2,3,4 or 5,with higher scores indicating greater disability.Negative change from Baseline(BL)indicates improvement.Change from BL in mFARS-neuro was analyzed using MMRM ANCOVA with BL as covariate;pooled site,visit,treatment,ambulation status as fixed factors;treatment-by-visit,BL mFARS-neuro-by visit interactions.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change at Week 2, Cough (0-2): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Cough (0-2) | 0.06 (0.051) | 0.07 (0.072) | 0.06 (0.051)
  Change at Week 7, Cough (0-2): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Cough (0-2) | 0.01 (0.063) | -0.05 (0.087) | 0.11 (0.065)
  Change at Week 12, Cough (0-2): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Cough (0-2) | 0.01 (0.063) | 0.08 (0.088) | 0.13 (0.063)
  Change at Week 2, Speech (0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Speech (0-3) | 0.00 (0.058) | 0.08 (0.083) | 0.10 (0.060)
  Change at Week 7, Speech (0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Speech (0-3) | 0.00 (0.043) | -0.04 (0.060) | 0.07 (0.045)
  Change at Week 12, Speech (0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Speech (0-3) | 0.00 (0.056) | 0.00 (0.079) | 0.09 (0.057)
  Change at Week 2,Right Finger to Finger Test(0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2,Right Finger to Finger Test(0-3) | 0.10 (0.079) | 0.17 (0.109) | 0.06 (0.078)
  Change at Week 7,Right Finger to Finger Test(0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7,Right Finger to Finger Test(0-3) | 0.04 (0.075) | 0.12 (0.102) | -0.02 (0.075)
  Change at Week 12,Right Finger to Finger Test(0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12,Right Finger to Finger Test(0-3) | 0.21 (0.077) | 0.12 (0.105) | 0.06 (0.074)
  Change at Week 2, Left Finger to Finger Test (0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Finger to Finger Test (0-3) | 0.04 (0.085) | 0.13 (0.120) | 0.07 (0.084)
  Change at Week 7, Left Finger to Finger Test (0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Left Finger to Finger Test (0-3) | 0.05 (0.075) | 0.07 (0.104) | 0.07 (0.077)
  Change at Week 12,Left Finger to Finger Test(0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12,Left Finger to Finger Test(0-3) | 0.13 (0.095) | 0.22 (0.132) | 0.04 (0.093)
  Change at Week 2, Right Nose to Finger Test (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Right Nose to Finger Test (0-4) | -0.08 (0.085) | 0.21 (0.126) | 0.06 (0.085)
  Change at Week 7, Right Nose to Finger Test (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Right Nose to Finger Test (0-4) | 0.01 (0.103) | 0.09 (0.147) | -0.07 (0.107)
  Change at Week 12, Right Nose to Finger Test (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Right Nose to Finger Test (0-4) | 0.00 (0.098) | -0.15 (0.140) | 0.00 (0.097)
  Change at Week 2, Left Nose to Finger Test (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Nose to Finger Test (0-4) | -0.05 (0.096) | 0.08 (0.137) | 0.05 (0.095)
  Change at Week 7, Left Nose to Finger Test (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Left Nose to Finger Test (0-4) | 0.15 (0.095) | 0.32 (0.133) | 0.01 (0.098)
  Change at Week 12, Left Nose to Finger Test (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Left Nose to Finger Test (0-4) | 0.11 (0.103) | 0.10 (0.141) | 0.14 (0.099)
  Change at Week 2, Right Dysmetria Test (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Right Dysmetria Test (0-4) | -0.11 (0.106) | -0.15 (0.151) | 0.01 (0.105)
  Change at Week 7, Right Dysmetria Test (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Right Dysmetria Test (0-4) | -0.23 (0.129) | -0.11 (0.181) | -0.06 (0.134)
  Change at Week 12, Right Dysmetria Test (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Right Dysmetria Test (0-4) | -0.11 (0.132) | 0.01 (0.185) | -0.16 (0.130)
  Change at Week 2, Left Dysmetria Test (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Dysmetria Test (0-4) | -0.27 (0.111) | 0.02 (0.160) | -0.12 (0.110)
  Change at Week 7, Left Dysmetria Test (0-4): number analyzed (Participants) | 27 | 13 | 23
  Change at Week 7, Left Dysmetria Test (0-4) | -0.02 (0.136) | -0.26 (0.191) | -0.16 (0.141)
  Change at Week 12, Left Dysmetria Test (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Left Dysmetria Test (0-4) | -0.17 (0.151) | -0.11 (0.211) | 0.06 (0.149)
  Change at Week 2, RAM of Right Hands (0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, RAM of Right Hands (0-3) | -0.18 (0.103) | 0.05 (0.145) | -0.06 (0.102)
  Change at Week 7, RAM of Right Hands (0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, RAM of Right Hands (0-3) | 0.03 (0.122) | -0.03 (0.170) | 0.03 (0.126)
  Change at Week 12, RAM of Right Hands (0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, RAM of Right Hands (0-3) | -0.07 (0.113) | 0.12 (0.156) | -0.12 (0.112)
  Change at Week 2, RAM of Left Hands (0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, RAM of Left Hands (0-3) | -0.11 (0.085) | -0.03 (0.120) | -0.03 (0.085)
  Change at Week 7, RAM of Left Hands (0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, RAM of Left Hands (0-3) | -0.08 (0.123) | 0.01 (0.173) | 0.05 (0.129)
  Change at Week 12, RAM of Left Hands (0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, RAM of Left Hands (0-3) | -0.20 (0.096) | 0.11 (0.133) | 0.02 (0.095)
  Change at Week 2, Right Finger Taps (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Right Finger Taps (0-4) | -0.39 (0.121) | 0.05 (0.172) | -0.23 (0.124)
  Change at Week 7, Right Finger Taps (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Right Finger Taps (0-4) | -0.18 (0.136) | 0.04 (0.190) | -0.19 (0.143)
  Change at Week 12, Right Finger Taps (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Right Finger Taps (0-4) | -0.31 (0.140) | -0.13 (0.195) | -0.37 (0.140)
  Change at Week 2, Left Finger Taps (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Finger Taps (0-4) | -0.22 (0.132) | 0.28 (0.189) | -0.17 (0.132)
  Change at Week 7, Left Finger Taps (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Left Finger Taps (0-4) | -0.37 (0.131) | 0.22 (0.182) | -0.21 (0.136)
  Change at Week 12, Left Finger Taps (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Left Finger Taps (0-4) | -0.50 (0.161) | 0.07 (0.225) | -0.17 (0.160)
  Change at Week 2,Right Heel Along Shin Slide(0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2,Right Heel Along Shin Slide(0-4) | -0.24 (0.118) | -0.04 (0.166) | -0.24 (0.117)
  Change at Week 7,Right Heel Along Shin Slide(0-4): number analyzed (Participants) | 25 | 13 | 23
  Change at Week 7,Right Heel Along Shin Slide(0-4) | -0.18 (0.152) | -0.32 (0.209) | -0.35 (0.155)
  Change at Week 12,Right Heel Along Shin Slide(0-4): number analyzed (Participants) | 23 | 12 | 24
  Change at Week 12,Right Heel Along Shin Slide(0-4) | -0.43 (0.164) | -0.09 (0.223) | -0.30 (0.160)
  Change at Week 2, Left Heel Along Shin Slide (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Heel Along Shin Slide (0-4) | 0.01 (0.121) | -0.15 (0.174) | 0.05 (0.121)
  Change at Week 7, Left Heel Along Shin Slide (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Left Heel Along Shin Slide (0-4) | 0.08 (0.133) | -0.23 (0.187) | -0.09 (0.138)
  Change at Week 12,Left Heel Along Shin Slide(0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12,Left Heel Along Shin Slide(0-4) | -0.16 (0.151) | -0.18 (0.210) | -0.15 (0.149)
  Change at Week 2, Right Heel Along Shin Tap (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Right Heel Along Shin Tap (0-4) | -0.39 (0.114) | -0.17 (0.159) | 0.04 (0.113)
  Change at Week 7, Right Heel Along Shin Tap (0-4): number analyzed (Participants) | 25 | 13 | 23
  Change at Week 7, Right Heel Along Shin Tap (0-4) | -0.14 (0.163) | -0.41 (0.224) | -0.14 (0.168)
  Change at Week 12, Right Heel Along Shin Tap (0-4): number analyzed (Participants) | 23 | 12 | 24
  Change at Week 12, Right Heel Along Shin Tap (0-4) | -0.32 (0.137) | -0.18 (0.184) | 0.01 (0.131)
  Change at Week 2, Left Heel Along Shin Tap (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Left Heel Along Shin Tap (0-4) | -0.38 (0.121) | -0.22 (0.171) | -0.05 (0.120)
  Change at Week 7, Left Heel Along Shin Tap (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Left Heel Along Shin Tap (0-4) | -0.36 (0.165) | 0.01 (0.230) | -0.15 (0.171)
  Change at Week 12, Left Heel Along Shin Tap (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Left Heel Along Shin Tap (0-4) | -0.52 (0.180) | -0.21 (0.251) | -0.27 (0.178)
  Change at Week 2, Siting Posture (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Siting Posture (0-4) | -0.3 (0.11) | -0.1 (0.15) | -0.1 (0.11)
  Change at Week 7, Siting Posture (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Siting Posture (0-4) | -0.4 (0.11) | -0.5 (0.15) | -0.2 (0.11)
  Change at Week 12, Siting Posture (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Siting Posture (0-4) | -0.1 (0.12) | -0.3 (0.16) | -0.1 (0.11)
  Change at Week 2, SFA -TTA (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, SFA -TTA (0-4) | -0.1 (0.15) | 0.0 (0.21) | -0.1 (0.15)
  Change at Week 7, SFA - TTA (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, SFA - TTA (0-4) | 0.1 (0.12) | 0.0 (0.17) | -0.1 (0.12)
  Change at Week 12, SFA - TTA (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, SFA - TTA (0-4) | -0.1 (0.13) | 0.0 (0.19) | 0.0 (0.13)
  Change at Week 2, SFA (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, SFA (Eyes Closed) - TTA (0-4) | 0.0 (0.07) | 0.1 (0.10) | -0.1 (0.07)
  Change at Week 7, SFA (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, SFA (Eyes Closed) - TTA (0-4) | 0.2 (0.11) | 0.1 (0.16) | 0.0 (0.12)
  Change at Week 12, SFA (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, SFA (Eyes Closed) - TTA (0-4) | 0.2 (0.14) | 0.2 (0.19) | 0.0 (0.14)
  Change at Week 2, SFT - TTA (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, SFT - TTA (0-4) | 0.0 (0.18) | -0.3 (0.26) | 0.4 (0.19)
  Change at Week 7, SFT - TTA (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, SFT - TTA (0-4) | -0.1 (0.11) | -0.1 (0.15) | 0.3 (0.11)
  Change at Week 12, SFT - TTA (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, SFT - TTA (0-4) | 0.0 (0.14) | -0.2 (0.19) | 0.3 (0.14)
  Change at Week 2, SFT (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, SFT (Eyes Closed) - TTA (0-4) | 0.1 (0.06) | 0.1 (0.09) | 0.0 (0.06)
  Change at Week 7, SFT (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, SFT (Eyes Closed) - TTA (0-4) | 0.1 (0.06) | 0.1 (0.09) | 0.1 (0.07)
  Change at Week 12, SFT (Eyes Closed) - TTA (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, SFT (Eyes Closed) - TTA (0-4) | 0.0 (0.07) | 0.0 (0.09) | -0.1 (0.06)
  Change at Week 2, Tandem Stance - TTA (0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Tandem Stance - TTA (0-4) | 0.0 (0.05) | 0.0 (0.07) | 0.0 (0.05)
  Change at Week 7, Tandem Stance - TTA (0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Tandem Stance - TTA (0-4) | 0.0 (0.05) | -0.1 (0.07) | 0.1 (0.05)
  Change at Week 12, Tandem Stance - TTA (0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Tandem Stance - TTA (0-4) | 0.1 (0.05) | 0.0 (0.07) | 0.1 (0.05)
  Change at Week 2,Stance on Dominant Foot-TTA(0-4): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2,Stance on Dominant Foot-TTA(0-4) | NA (NA) — The least squares (LS) mean and standard error (SE) was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point.
  Change at Week 7,Stance on Dominant Foot-TTA(0-4): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7,Stance on Dominant Foot-TTA(0-4) | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point.
  Change at Week 12,Stance on Dominant Foot-TTA(0-4): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12,Stance on Dominant Foot-TTA(0-4) | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point. | NA (NA) — The LS mean and SE was not estimable as there was no change from baseline in subscale score at this time point.
  Change at Week 2, Tandem Walk (0-3): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Tandem Walk (0-3) | 0.0 (0.05) | 0.0 (0.07) | 0.0 (0.05)
  Change at Week 7, Tandem Walk (0-3): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Tandem Walk (0-3) | 0.0 (0.05) | -0.1 (0.07) | 0.0 (0.05)
  Change at Week 12, Tandem Walk (0-3): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Tandem Walk (0-3) | 0.0 (0.06) | -0.1 (0.08) | 0.0 (0.06)
  Change at Week 2, Gait (0-5): number analyzed (Participants) | 27 | 13 | 26
  Change at Week 2, Gait (0-5) | -0.3 (0.12) | -0.2 (0.17) | 0.2 (0.12)
  Change at Week 7, Gait (0-5): number analyzed (Participants) | 26 | 13 | 23
  Change at Week 7, Gait (0-5) | -0.1 (0.11) | -0.3 (0.15) | 0.2 (0.11)
  Change at Week 12, Gait (0-5): number analyzed (Participants) | 24 | 12 | 24
  Change at Week 12, Gait (0-5) | -0.1 (0.11) | -0.2 (0.15) | 0.1 (0.10)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Cough; Test type: Superiority; Least Squares Mean Difference = 0.01, 90% CI 2-sided [-0.13 to 0.15], Standard Error of Mean 0.084
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Cough; Test type: Superiority; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.11 to 0.12], Standard Error of Mean 0.069
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Cough; Test type: Superiority; Least Squares Mean Difference = -0.06, 90% CI 2-sided [-0.24 to 0.11], Standard Error of Mean 0.105
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Cough; Test type: Superiority; Least Squares Mean Difference = 0.10, 90% CI 2-sided [-0.05 to 0.25], Standard Error of Mean 0.088
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Cough; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.11 to 0.25], Standard Error of Mean 0.106
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Cough; Test type: Superiority; Least Squares Mean Difference = 0.12, 90% CI 2-sided [-0.03 to 0.26], Standard Error of Mean 0.087
Statistical Analysis 7: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Speech; Test type: Superiority; Least Squares Mean Difference = 0.08, 90% CI 2-sided [-0.09 to 0.25], Standard Error of Mean 0.100
Statistical Analysis 8: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Speech; Test type: Superiority; Least Squares Mean Difference = 0.10, 90% CI 2-sided [-0.04 to 0.24], Standard Error of Mean 0.083
Statistical Analysis 9: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Speech; Test type: Superiority; Least Squares Mean Difference = -0.04, 90% CI 2-sided [-0.16 to 0.08], Standard Error of Mean 0.071
Statistical Analysis 10: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Speech; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.03 to 0.17], Standard Error of Mean 0.060
Statistical Analysis 11: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Speech; Test type: Superiority; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.16 to 0.16], Standard Error of Mean 0.095
Statistical Analysis 12: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Speech; Test type: Superiority; Least Squares Mean Difference = 0.09, 90% CI 2-sided [-0.04 to 0.22], Standard Error of Mean 0.079
Statistical Analysis 13: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.14 to 0.29], Standard Error of Mean 0.131
Statistical Analysis 14: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.04, 90% CI 2-sided [-0.22 to 0.14], Standard Error of Mean 0.108
Statistical Analysis 15: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.13 to 0.28], Standard Error of Mean 0.122
Statistical Analysis 16: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.07, 90% CI 2-sided [-0.24 to 0.11], Standard Error of Mean 0.103
Statistical Analysis 17: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.09, 90% CI 2-sided [-0.30 to 0.12], Standard Error of Mean 0.126
Statistical Analysis 18: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Right Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.14, 90% CI 2-sided [-0.32 to 0.03], Standard Error of Mean 0.104
Statistical Analysis 19: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.09, 90% CI 2-sided [-0.15 to 0.33], Standard Error of Mean 0.142
Statistical Analysis 20: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.04, 90% CI 2-sided [-0.16 to 0.23], Standard Error of Mean 0.117
Statistical Analysis 21: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.03, 90% CI 2-sided [-0.18 to 0.23], Standard Error of Mean 0.123
Statistical Analysis 22: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.03, 90% CI 2-sided [-0.15 to 0.20], Standard Error of Mean 0.104
Statistical Analysis 23: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.09, 90% CI 2-sided [-0.17 to 0.36], Standard Error of Mean 0.158
Statistical Analysis 24: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Finger to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.09, 90% CI 2-sided [-0.30 to 0.13], Standard Error of Mean 0.130
Statistical Analysis 25: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.29, 90% CI 2-sided [0.04 to 0.53], Standard Error of Mean 0.145
Statistical Analysis 26: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.14, 90% CI 2-sided [-0.06 to 0.33], Standard Error of Mean 0.118
Statistical Analysis 27: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.07, 90% CI 2-sided [-0.22 to 0.37], Standard Error of Mean 0.174
Statistical Analysis 28: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.08, 90% CI 2-sided [-0.32 to 0.16], Standard Error of Mean 0.146
Statistical Analysis 29: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.15, 90% CI 2-sided [-0.43 to 0.12], Standard Error of Mean 0.166
Statistical Analysis 30: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Right Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.23 to 0.23], Standard Error of Mean 0.136
Statistical Analysis 31: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.13, 90% CI 2-sided [-0.14 to 0.40], Standard Error of Mean 0.161
Statistical Analysis 32: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.10, 90% CI 2-sided [-0.12 to 0.33], Standard Error of Mean 0.133
Statistical Analysis 33: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.17, 90% CI 2-sided [-0.09 to 0.43], Standard Error of Mean 0.157
Statistical Analysis 34: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.13, 90% CI 2-sided [-0.36 to 0.09], Standard Error of Mean 0.134
Statistical Analysis 35: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = -0.01, 90% CI 2-sided [-0.29 to 0.27], Standard Error of Mean 0.169
Statistical Analysis 36: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Nose to Finger Test; Test type: Superiority; Least Squares Mean Difference = 0.03, 90% CI 2-sided [-0.21 to 0.27], Standard Error of Mean 0.141
Statistical Analysis 37: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = -0.04, 90% CI 2-sided [-0.33 to 0.26], Standard Error of Mean 0.176
Statistical Analysis 38: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.12, 90% CI 2-sided [-0.12 to 0.36], Standard Error of Mean 0.145
Statistical Analysis 39: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.12, 90% CI 2-sided [-0.25 to 0.48], Standard Error of Mean 0.217
Statistical Analysis 40: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.17, 90% CI 2-sided [-0.14 to 0.47], Standard Error of Mean 0.183
Statistical Analysis 41: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.11, 90% CI 2-sided [-0.26 to 0.48], Standard Error of Mean 0.221
Statistical Analysis 42: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Right Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = -0.06, 90% CI 2-sided [-0.36 to 0.25], Standard Error of Mean 0.183
Statistical Analysis 43: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.29, 90% CI 2-sided [-0.02 to 0.60], Standard Error of Mean 0.185
Statistical Analysis 44: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.15, 90% CI 2-sided [-0.10 to 0.41], Standard Error of Mean 0.153
Statistical Analysis 45: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = -0.25, 90% CI 2-sided [-0.63 to 0.13], Standard Error of Mean 0.228
Statistical Analysis 46: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = -0.14, 90% CI 2-sided [-0.47 to 0.18], Standard Error of Mean 0.192
Statistical Analysis 47: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.06, 90% CI 2-sided [-0.37 to 0.48], Standard Error of Mean 0.254
Statistical Analysis 48: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Dysmetria Test; Test type: Superiority; Least Squares Mean Difference = 0.23, 90% CI 2-sided [-0.11 to 0.58], Standard Error of Mean 0.209
Statistical Analysis 49: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = 0.22, 90% CI 2-sided [-0.06 to 0.51], Standard Error of Mean 0.170
Statistical Analysis 50: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = 0.11, 90% CI 2-sided [-0.12 to 0.35], Standard Error of Mean 0.141
Statistical Analysis 51: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = -0.06, 90% CI 2-sided [-0.41 to 0.28], Standard Error of Mean 0.204
Statistical Analysis 52: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.29 to 0.29], Standard Error of Mean 0.172
Statistical Analysis 53: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = 0.19, 90% CI 2-sided [-0.12 to 0.51], Standard Error of Mean 0.187
Statistical Analysis 54: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, RAM of Right Hands; Test type: Superiority; Least Squares Mean Difference = -0.05, 90% CI 2-sided [-0.31 to 0.21], Standard Error of Mean 0.156
Statistical Analysis 55: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, RAM of Left Hands; Test type: Superiority; Least Squares Mean Difference = 0.08, 90% CI 2-sided [-0.15 to 0.32], Standard Error of Mean 0.141
Statistical Analysis 56: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, RAM of Left Hands; Test type: Superiority; Least Squares Mean Difference = 0.08, 90% CI 2-sided [-0.12 to 0.27], Standard Error of Mean 0.116
Statistical Analysis 57: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, RAM of Left Hands; Test type: Superiority; Least Squares Mean Difference = 0.08, 90% CI 2-sided [-0.27 to 0.43], Standard Error of Mean 0.209
Statistical Analysis 58: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, RAM of Left Hands; Test type: Superiority; Least Squares Mean Difference = 0.12, 90% CI 2-sided [-0.17 to 0.42], Standard Error of Mean 0.176
Statistical Analysis 59: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, RAM of Left Hand; Test type: Superiority; Least Squares Mean Difference = 0.31, 90% CI 2-sided [0.04 to 0.58], Standard Error of Mean 0.159
Statistical Analysis 60: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, RAM of Left Hand; Test type: Superiority; Least Squares Mean Difference = 0.21, 90% CI 2-sided [-0.01 to 0.43], Standard Error of Mean 0.132
Statistical Analysis 61: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.44, 90% CI 2-sided [0.10 to 0.77], Standard Error of Mean 0.201
Statistical Analysis 62: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-0.12 to 0.44], Standard Error of Mean 0.168
Statistical Analysis 63: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.22, 90% CI 2-sided [-0.16 to 0.60], Standard Error of Mean 0.227
Statistical Analysis 64: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = -0.01, 90% CI 2-sided [-0.33 to 0.31], Standard Error of Mean 0.193
Statistical Analysis 65: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.17, 90% CI 2-sided [-0.22 to 0.56], Standard Error of Mean 0.233
Statistical Analysis 66: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Right Finger Taps; Test type: Superiority; Least Squares Mean Difference = -0.07, 90% CI 2-sided [-0.39 to 0.26], Standard Error of Mean 0.194
Statistical Analysis 67: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.50, 90% CI 2-sided [0.12 to 0.87], Standard Error of Mean 0.223
Statistical Analysis 68: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.05, 90% CI 2-sided [-0.25 to 0.36], Standard Error of Mean 0.183
Statistical Analysis 69: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.59, 90% CI 2-sided [0.22 to 0.95], Standard Error of Mean 0.218
Statistical Analysis 70: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-0.15 to 0.47], Standard Error of Mean 0.184
Statistical Analysis 71: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.57, 90% CI 2-sided [0.11 to 1.02], Standard Error of Mean 0.272
Statistical Analysis 72: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Finger Taps; Test type: Superiority; Least Squares Mean Difference = 0.33, 90% CI 2-sided [-0.04 to 0.71], Standard Error of Mean 0.224
Statistical Analysis 73: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.20, 90% CI 2-sided [-0.12 to 0.53], Standard Error of Mean 0.193
Statistical Analysis 74: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.01, 90% CI 2-sided [-0.26 to 0.27], Standard Error of Mean 0.161
Statistical Analysis 75: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.14, 90% CI 2-sided [-0.56 to 0.28], Standard Error of Mean 0.251
Statistical Analysis 76: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.17, 90% CI 2-sided [-0.53 to 0.19], Standard Error of Mean 0.214
Statistical Analysis 77: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12,Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.33, 90% CI 2-sided [-0.12 to 0.78], Standard Error of Mean 0.270
Statistical Analysis 78: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12,Right Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.13, 90% CI 2-sided [-0.25 to 0.51], Standard Error of Mean 0.226
Statistical Analysis 79: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.17, 90% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.205
Statistical Analysis 80: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.03, 90% CI 2-sided [-0.25 to 0.31], Standard Error of Mean 0.166
Statistical Analysis 81: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.31, 90% CI 2-sided [-0.68 to 0.07], Standard Error of Mean 0.224
Statistical Analysis 82: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.17, 90% CI 2-sided [-0.48 to 0.15], Standard Error of Mean 0.188
Statistical Analysis 83: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = -0.02, 90% CI 2-sided [-0.45 to 0.40], Standard Error of Mean 0.254
Statistical Analysis 84: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Heel Along Shin Slide; Test type: Superiority; Least Squares Mean Difference = 0.01, 90% CI 2-sided [-0.34 to 0.36], Standard Error of Mean 0.209
Statistical Analysis 85: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.22, 90% CI 2-sided [-0.10 to 0.53], Standard Error of Mean 0.187
Statistical Analysis 86: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.43, 90% CI 2-sided [0.17 to 0.69], Standard Error of Mean 0.155
Statistical Analysis 87: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = -0.27, 90% CI 2-sided [-0.72 to 0.19], Standard Error of Mean 0.272
Statistical Analysis 88: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.00, 90% CI 2-sided [-0.38 to 0.39], Standard Error of Mean 0.231
Statistical Analysis 89: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.14, 90% CI 2-sided [-0.23 to 0.51], Standard Error of Mean 0.222
Statistical Analysis 90: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Right Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.33, 90% CI 2-sided [0.02 to 0.64], Standard Error of Mean 0.186
Statistical Analysis 91: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-0.17 to 0.50], Standard Error of Mean 0.199
Statistical Analysis 92: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.34, 90% CI 2-sided [0.06 to 0.61], Standard Error of Mean 0.164
Statistical Analysis 93: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.37, 90% CI 2-sided [-0.09 to 0.84], Standard Error of Mean 0.277
Statistical Analysis 94: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.21, 90% CI 2-sided [-0.19 to 0.60], Standard Error of Mean 0.234
Statistical Analysis 95: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.31, 90% CI 2-sided [-0.20 to 0.82], Standard Error of Mean 0.303
Statistical Analysis 96: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Left Heel Along Shin Tap; Test type: Superiority; Least Squares Mean Difference = 0.25, 90% CI 2-sided [-0.17 to 0.67], Standard Error of Mean 0.250
Statistical Analysis 97: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Siting Posture; Test type: Superiority; Least Squares Mean Difference = 0.2, 90% CI 2-sided [-0.1 to 0.5], Standard Error of Mean 0.18
Statistical Analysis 98: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Siting Posture; Test type: Superiority; Least Squares Mean Difference = 0.2, 90% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.15
Statistical Analysis 99: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Siting Posture; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.18
Statistical Analysis 100: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Siting Posture; Test type: Superiority; Least Squares Mean Difference = 0.2, 90% CI 2-sided [0.0 to 0.5], Standard Error of Mean 0.15
Statistical Analysis 101: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Siting Posture; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.19
Statistical Analysis 102: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Siting Posture; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.16
Statistical Analysis 103: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.25
Statistical Analysis 104: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.20
Statistical Analysis 105: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.20
Statistical Analysis 106: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.17
Statistical Analysis 107: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.22
Statistical Analysis 108: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, SFA - TTA; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.19
Statistical Analysis 109: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.11
Statistical Analysis 110: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 111: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.19
Statistical Analysis 112: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.16
Statistical Analysis 113: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.23
Statistical Analysis 114: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, SFA (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.19
Statistical Analysis 115: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = -0.3, 90% CI 2-sided [-0.8 to 0.2], Standard Error of Mean 0.32
Statistical Analysis 116: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = 0.4, 90% CI 2-sided [0.0 to 0.8], Standard Error of Mean 0.26
Statistical Analysis 117: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.18
Statistical Analysis 118: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = 0.4, 90% CI 2-sided [0.2 to 0.7], Standard Error of Mean 0.15
Statistical Analysis 119: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.23
Statistical Analysis 120: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, SFT - TTA; Test type: Superiority; Least Squares Mean Difference = 0.3, 90% CI 2-sided [0.0 to 0.7], Standard Error of Mean 0.19
Statistical Analysis 121: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.11
Statistical Analysis 122: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 123: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 124: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 125: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 126: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, SFT (Eyes Closed) - TTA; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 127: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 128: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 129: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 130: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.07
Statistical Analysis 131: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 132: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Tandem Stance - TTA; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.07
Statistical Analysis 133: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 134: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 135: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 136: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 137: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.10
Statistical Analysis 138: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Tandem Walk; Test type: Superiority; Least Squares Mean Difference = 0.0, 90% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 139: Comparison: Placebo vs TAK-831 75 mg; Change at Week 2, Gait; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.20
Statistical Analysis 140: Comparison: Placebo vs TAK-831 300 mg; Change at Week 2, Gait; Test type: Superiority; Least Squares Mean Difference = 0.4, 90% CI 2-sided [0.1 to 0.7], Standard Error of Mean 0.17
Statistical Analysis 141: Comparison: Placebo vs TAK-831 75 mg; Change at Week 7, Gait; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.17
Statistical Analysis 142: Comparison: Placebo vs TAK-831 300 mg; Change at Week 7, Gait; Test type: Superiority; Least Squares Mean Difference = 0.3, 90% CI 2-sided [0.1 to 0.6], Standard Error of Mean 0.15
Statistical Analysis 143: Comparison: Placebo vs TAK-831 75 mg; Change at Week 12, Gait; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.17
Statistical Analysis 144: Comparison: Placebo vs TAK-831 300 mg; Change at Week 12, Gait; Test type: Superiority; Least Squares Mean Difference = 0.3, 90% CI 2-sided [0.0 to 0.5], Standard Error of Mean 0.14

8. Secondary Outcome: Change From Baseline in the Timed 25-Foot Walk (T25FW)
Description: The participant was instructed to walk 25 feet as quickly as possible, but safely. The time was calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task was immediately administered again by having the participant walk back the same distance. The two trials were averaged. A negative change from Baseline indicates improvement. Change from Baseline in T25FW was analyzed using MMRM ANCOVA with Baseline T25FW as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline T25FW-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
seconds
  Change from Baseline at Week 2: number analyzed (Participants) | 11 | 6 | 12
  Change from Baseline at Week 2 | 0.61 (0.901) | 0.84 (1.124) | 1.95 (0.990)
  Change from Baseline at Week 7: number analyzed (Participants) | 11 | 6 | 11
  Change from Baseline at Week 7 | 1.67 (0.948) | 1.77 (1.255) | 1.37 (1.080)
  Change from Baseline at Week 12: number analyzed (Participants) | 11 | 5 | 10
  Change from Baseline at Week 12 | 0.52 (0.903) | 2.70 (1.226) | 1.30 (1.057)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.599, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.23, 90% CI 2-sided [-1.31 to 1.76], Standard Error of Mean 0.889
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.978, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 1.34, 90% CI 2-sided [0.26 to 2.42], Standard Error of Mean 0.625
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.533, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.09, 90% CI 2-sided [-1.87 to 2.06], Standard Error of Mean 1.140
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.370, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.30, 90% CI 2-sided [-1.83 to 1.23], Standard Error of Mean 0.886
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.972, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 2.18, 90% CI 2-sided [0.32 to 4.04], Standard Error of Mean 1.078
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.825, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.78, 90% CI 2-sided [-0.63 to 2.19], Standard Error of Mean 0.819

9. Secondary Outcome: Change From Baseline in the 9-HPT and T25FW Composite Score
Description: 9-HPT and T25FW were evaluated together as a performance-based composite measure. The inverse transform of each score was computed. The inverse scores from each test were tabulated and converted to test-specific Z scores by subtracting the cohort mean from the raw score, and then dividing by the cohort standard deviation (SD) to create a Z score for the test. The composite Z scores were created by subtracting Z-score for T25FW from the Z-score for 9-HPT-1. A larger Z-score represents a better outcome. A positive change from Baseline indicates improvement. Change from Baseline in composite score was analyzed using MMRM ANCOVA with Baseline composite score as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline composite score-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
z-score
  Change from Baseline at Week 2: number analyzed (Participants) | 11 | 6 | 12
  Change from Baseline at Week 2 | 0.1369 (0.21905) | 0.1819 (0.28555) | -0.1911 (0.24051)
  Change from Baseline at Week 7: number analyzed (Participants) | 11 | 6 | 11
  Change from Baseline at Week 7 | -0.1112 (0.24167) | 0.0336 (0.32731) | -0.0998 (0.26792)
  Change from Baseline at Week 12: number analyzed (Participants) | 11 | 5 | 10
  Change from Baseline at Week 12 | 0.0060 (0.22484) | -0.2007 (0.31057) | 0.1233 (0.25501)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.426, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.0450, 90% CI 2-sided [-0.3665 to 0.4565], Standard Error of Mean 0.23858
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.975, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.3281, 90% CI 2-sided [-0.6005 to -0.0557], Standard Error of Mean 0.15794
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.324, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.1448, 90% CI 2-sided [-0.3931 to 0.6826], Standard Error of Mean 0.31186
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.481, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.0113, 90% CI 2-sided [-0.3891 to 0.4117], Standard Error of Mean 0.23213
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.765, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.2067, 90% CI 2-sided [-0.6911 to 0.2778], Standard Error of Mean 0.28088
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.280, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.1173, 90% CI 2-sided [-0.2238 to 0.4585], Standard Error of Mean 0.19778

10. Secondary Outcome: Change From Baseline in Low-Contrast Letter Acuity (LCLA) Test Score
Description: The LCLA test assessed visual function in both eyes using the Low-Contrast Sloan Letter Charts at different contrast levels. The score ranged from 0 to 70, where 0=worst visual functioning and 70=best visual functioning. A positive change from Baseline indicates improvement. The change from Baseline in LCLA was analyzed using MMRM ANCOVA with Baseline LCLA as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline LCLA-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7, and, 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 27 | 13 | 26
  Change from Baseline at Week 2 | 1.8 (2.56) | -0.9 (3.61) | 5.1 (2.53)
  Change from Baseline at Week 7: number analyzed (Participants) | 26 | 13 | 24
  Change from Baseline at Week 7 | 4.6 (2.20) | -2.3 (3.06) | 6.0 (2.17)
  Change from Baseline at Week 12: number analyzed (Participants) | 24 | 12 | 24
  Change from Baseline at Week 12 | 0.0 (2.61) | -5.7 (3.65) | 3.1 (2.56)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.735, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.7, 90% CI 2-sided [-9.9 to 4.4], Standard Error of Mean 4.28
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.182, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 3.2, 90% CI 2-sided [-2.7 to 9.1], Standard Error of Mean 3.51
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.970, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -6.9, 90% CI 2-sided [-12.9 to -0.9], Standard Error of Mean 3.59
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.321, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 1.4, 90% CI 2-sided [-3.6 to 6.4], Standard Error of Mean 3.00
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.905, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -5.8, 90% CI 2-sided [-13.0 to 1.5], Standard Error of Mean 4.34
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.199, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 3.1, 90% CI 2-sided [-2.9 to 9.0], Standard Error of Mean 3.57

11. Secondary Outcome: Number of Participants by Clinical Global Impression-Improvement (CGI-I) (Global Change) Score Categories
Description: The clinician used the CGI-I scale to assess the participant's improvement (or worsening) overall relative to Baseline on a 7-point scale where: 1=Much improved, 2=Moderately improved, 3=A little improved, 4=No change, 5=A little worse, 6=Moderately worse and 7=Much worse. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Week 2, Moderately Improved: number analyzed (Participants) | 27 | 13 | 25
  Week 2, Moderately Improved | 1 | 0 | 2
  Week 2, A Little Improved: number analyzed (Participants) | 27 | 13 | 25
  Week 2, A Little Improved | 14 | 3 | 6
  Week 2, No Change: number analyzed (Participants) | 27 | 13 | 25
  Week 2, No Change | 11 | 10 | 17
  Week 2, A little Worse: number analyzed (Participants) | 27 | 13 | 25
  Week 2, A little Worse | 1 | 0 | 0
  Week 7, Moderately Improved: number analyzed (Participants) | 26 | 13 | 21
  Week 7, Moderately Improved | 1 | 0 | 1
  Week 7, A Little Improved: number analyzed (Participants) | 26 | 13 | 21
  Week 7, A Little Improved | 13 | 4 | 8
  Week 7, No Change: number analyzed (Participants) | 26 | 13 | 21
  Week 7, No Change | 11 | 8 | 11
  Week 7, A little Worse: number analyzed (Participants) | 26 | 13 | 21
  Week 7, A little Worse | 1 | 1 | 1
  Week 12, Moderately Improved: number analyzed (Participants) | 24 | 11 | 24
  Week 12, Moderately Improved | 1 | 0 | 0
  Week 12, A Little Improved: number analyzed (Participants) | 24 | 11 | 24
  Week 12, A Little Improved | 9 | 3 | 7
  Week 12, No Change: number analyzed (Participants) | 24 | 11 | 24
  Week 12, No Change | 12 | 7 | 16
  Week 12, A little Worse: number analyzed (Participants) | 24 | 11 | 24
  Week 12, A little Worse | 2 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.974, Cochran-Mantel-Haenszel — The p-value was obtained using the Cochran-Mantel-Haenszel row mean score test stratified by ambulation status at randomization
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.893, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.954, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.793, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.845, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.816, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Number of Participants by Patient Global Impression-Improvement (PGI-I) (Global Change) Score Categories
Description: The participant used the PGI-I scale to assess their improvement (or worsening) overall relative to Baseline on a 7-point scale where: 1=Much improved, 2=Moderately improved, 3=A little improved, 4=No change, 5=A little worse, 6=Moderately worse and 7=Much worse. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Weeks 2, 7 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Week 2, Moderately Improved: number analyzed (Participants) | 27 | 13 | 26
  Week 2, Moderately Improved | 2 | 0 | 0
  Week 2, A Little Improved: number analyzed (Participants) | 27 | 13 | 26
  Week 2, A Little Improved | 6 | 3 | 8
  Week 2, No Change: number analyzed (Participants) | 27 | 13 | 26
  Week 2, No Change | 19 | 10 | 16
  Week 2, A little Worse: number analyzed (Participants) | 27 | 13 | 26
  Week 2, A little Worse | 0 | 0 | 2
  Week 7, Moderately Improved: number analyzed (Participants) | 26 | 13 | 24
  Week 7, Moderately Improved | 3 | 0 | 3
  Week 7, A Little Improved: number analyzed (Participants) | 26 | 13 | 24
  Week 7, A Little Improved | 10 | 4 | 5
  Week 7, No Change: number analyzed (Participants) | 26 | 13 | 24
  Week 7, No Change | 11 | 8 | 14
  Week 7, A little Worse: number analyzed (Participants) | 26 | 13 | 24
  Week 7, A little Worse | 2 | 1 | 2
  Week 12, Much Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, Much Improved | 1 | 0 | 0
  Week 12, Moderately Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, Moderately Improved | 5 | 1 | 1
  Week 12, A Little Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, A Little Improved | 8 | 4 | 3
  Week 12, No Change: number analyzed (Participants) | 24 | 12 | 24
  Week 12, No Change | 7 | 7 | 15
  Week 12, A little Worse: number analyzed (Participants) | 24 | 12 | 24
  Week 12, A little Worse | 3 | 0 | 4
  Week 12, Moderately Worse: number analyzed (Participants) | 24 | 12 | 24
  Week 12, Moderately Worse | 0 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.840, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.854, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.922, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.794, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.830, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.998, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

13. Secondary Outcome: Number of Participants by CGI-I (Upper Extremity Functional Change) Score Categories
Description: The clinician used the CGI-I scale to assess the participant's improvement (or worsening) in upper extremity function relative to Baseline on a 7-point scale where: 1=Much improved, 2=Moderately improved, 3=A little improved, 4=No change, 5=A little worse, 6=Moderately worse and 7=Much worse. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Week 2, Moderately Improved: number analyzed (Participants) | 27 | 13 | 25
  Week 2, Moderately Improved | 1 | 0 | 2
  Week 2, A Little Improved: number analyzed (Participants) | 27 | 13 | 25
  Week 2, A Little Improved | 13 | 2 | 7
  Week 2, No Change: number analyzed (Participants) | 27 | 13 | 25
  Week 2, No Change | 12 | 11 | 16
  Week 2, A little Worse: number analyzed (Participants) | 27 | 13 | 25
  Week 2, A little Worse | 1 | 0 | 0
  Week 7, Moderately Improved: number analyzed (Participants) | 26 | 13 | 21
  Week 7, Moderately Improved | 1 | 1 | 0
  Week 7, A Little Improved: number analyzed (Participants) | 26 | 13 | 21
  Week 7, A Little Improved | 10 | 5 | 11
  Week 7, No Change: number analyzed (Participants) | 26 | 13 | 21
  Week 7, No Change | 14 | 6 | 7
  Week 7, A little Worse: number analyzed (Participants) | 26 | 13 | 21
  Week 7, A little Worse | 1 | 1 | 3
  Week 12, Moderately Improved: number analyzed (Participants) | 24 | 11 | 24
  Week 12, Moderately Improved | 2 | 2 | 0
  Week 12, A Little Improved: number analyzed (Participants) | 24 | 11 | 24
  Week 12, A Little Improved | 11 | 2 | 9
  Week 12, No Change: number analyzed (Participants) | 24 | 11 | 24
  Week 12, No Change | 9 | 7 | 15
  Week 12, A little Worse: number analyzed (Participants) | 24 | 11 | 24
  Week 12, A little Worse | 2 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.987, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.771, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.526, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.665, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.576, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.865, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

14. Secondary Outcome: Number of Participants by PGI-I (Upper Extremity Functional Change) Score Categories
Description: The participant used the PGI-I scale to assess their improvement (or worsening) in upper extremity function relative to Baseline on a 7-point scale where: 1=Much improved, 2=Moderately improved, 3=A little improved, 4=No change, 5=A little worse, 6=Moderately worse and 7=Much worse. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Week 2, Moderately Improved: number analyzed (Participants) | 27 | 13 | 26
  Week 2, Moderately Improved | 5 | 0 | 0
  Week 2, A Little Improved: number analyzed (Participants) | 27 | 13 | 26
  Week 2, A Little Improved | 6 | 3 | 7
  Week 2, No Change: number analyzed (Participants) | 27 | 13 | 26
  Week 2, No Change | 16 | 10 | 18
  Week 2, A little Worse: number analyzed (Participants) | 27 | 13 | 26
  Week 2, A little Worse | 0 | 0 | 1
  Week 7, Much Improved: number analyzed (Participants) | 26 | 13 | 24
  Week 7, Much Improved | 0 | 0 | 1
  Week 7, Moderately Improved: number analyzed (Participants) | 26 | 13 | 24
  Week 7, Moderately Improved | 3 | 0 | 2
  Week 7, A Little Improved: number analyzed (Participants) | 26 | 13 | 24
  Week 7, A Little Improved | 10 | 4 | 4
  Week 7, No Change: number analyzed (Participants) | 26 | 13 | 24
  Week 7, No Change | 11 | 7 | 15
  Week 7, A little Worse: number analyzed (Participants) | 26 | 13 | 24
  Week 7, A little Worse | 2 | 2 | 2
  Week 12, Much Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, Much Improved | 2 | 0 | 0
  Week 12, Moderately Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, Moderately Improved | 6 | 1 | 1
  Week 12, A Little Improved: number analyzed (Participants) | 24 | 12 | 24
  Week 12, A Little Improved | 6 | 4 | 6
  Week 12, No Change: number analyzed (Participants) | 24 | 12 | 24
  Week 12, No Change | 9 | 7 | 15
  Week 12, A little Worse: number analyzed (Participants) | 24 | 12 | 24
  Week 12, A little Worse | 1 | 0 | 2
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.966, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.983, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.953, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.781, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.948, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.998, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

15. Secondary Outcome: Number of Participants by Clinical Global Impression-Severity (CGI-S) (Global Severity) Score Categories Relative to Baseline
Description: The clinician used the CGI-S scale to assess the severity of the participant's disease overall on a 5-point scale where: 0=No symptoms, 1=Mild, 2=Moderate, 3=Severe and 4=Very severe. The number of participants by CGI-S score category is reported relative to their CGI-S score at Baseline. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Score at Week 2=1 (Mild): number analyzed (Participants) | 6 | 4 | 3
  Score at Week 2=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=1 (Mild): Score at Baseline=1 (Mild) | 2 | 2 | 1
  Score at Week 2=1 (Mild): Score at Baseline=2 (Moderate) | 4 | 2 | 2
  Score at Week 2=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 | 0
  Score at Week 2=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=2 (Moderate): number analyzed (Participants) | 17 | 6 | 13
  Score at Week 2=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=2 (Moderate): Score at Baseline=1 (Mild) | 1 | 0 | 2
  Score at Week 2=2 (Moderate): Score at Baseline=2 (Moderate) | 14 | 6 | 10
  Score at Week 2=2 (Moderate): Score at Baseline=3 (Severe) | 2 | 0 | 1
  Score at Week 2=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=3 (Severe): number analyzed (Participants) | 3 | 2 | 9
  Score at Week 2=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 0
  Score at Week 2=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 0 | 1
  Score at Week 2=3 (Severe): Score at Baseline=3 (Severe) | 3 | 2 | 8
  Score at Week 2=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=4 (Very Severe): number analyzed (Participants) | 1 | 1 | 0
  Score at Week 2=4 (Very Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 |
  Score at Week 2=4 (Very Severe): Score at Baseline=1 (Mild) | 0 | 0 |
  Score at Week 2=4 (Very Severe): Score at Baseline=2 (Moderate) | 0 | 0 |
  Score at Week 2=4 (Very Severe): Score at Baseline=3 (Severe) | 0 | 0 |
  Score at Week 2=4 (Very Severe): Score at Baseline=4 (Very Severe) | 1 | 1 |
  Score at Week 7=1 (Mild): number analyzed (Participants) | 5 | 1 | 0
  Score at Week 7=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 |
  Score at Week 7=1 (Mild): Score at Baseline=1 (Mild) | 2 | 1 |
  Score at Week 7=1 (Mild): Score at Baseline=2 (Moderate) | 3 | 0 |
  Score at Week 7=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 |
  Score at Week 7=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 |
  Score at Week 7=2 (Moderate): number analyzed (Participants) | 18 | 10 | 16
  Score at Week 7=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 7=2 (Moderate): Score at Baseline=1 (Mild) | 1 | 1 | 3
  Score at Week 7=2 (Moderate): Score at Baseline=2 (Moderate) | 14 | 8 | 11
  Score at Week 7=2 (Moderate): Score at Baseline=3 (Severe) | 3 | 1 | 2
  Score at Week 7=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 7=3 (Severe): number analyzed (Participants) | 2 | 1 | 7
  Score at Week 7=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 7=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 0
  Score at Week 7=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 0 | 0
  Score at Week 7=3 (Severe): Score at Baseline=3 (Severe) | 2 | 1 | 7
  Score at Week 7=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 7=4 (Very Severe): number analyzed (Participants) | 1 | 1 | 0
  Score at Week 7=4 (Very Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 |
  Score at Week 7=4 (Very Severe): Score at Baseline=1 (Mild) | 0 | 0 |
  Score at Week 7=4 (Very Severe): Score at Baseline=2 (Moderate) | 0 | 0 |
  Score at Week 7=4 (Very Severe): Score at Baseline=3 (Severe) | 0 | 0 |
  Score at Week 7=4 (Very Severe): Score at Baseline=4 (Very Severe) | 1 | 1 |
  Score at Week 12=1 (Mild): number analyzed (Participants) | 6 | 1 | 3
  Score at Week 12=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=1 (Mild): Score at Baseline=1 (Mild) | 2 | 1 | 2
  Score at Week 12=1 (Mild): Score at Baseline=2 (Moderate) | 4 | 0 | 1
  Score at Week 12=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 | 0
  Score at Week 12=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=2 (Moderate): number analyzed (Participants) | 16 | 8 | 11
  Score at Week 12=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=2 (Moderate): Score at Baseline=1 (Mild) | 1 | 0 | 0
  Score at Week 12=2 (Moderate): Score at Baseline=2 (Moderate) | 13 | 8 | 11
  Score at Week 12=2 (Moderate): Score at Baseline=3 (Severe) | 2 | 0 | 0
  Score at Week 12=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=3 (Severe): number analyzed (Participants) | 1 | 1 | 10
  Score at Week 12=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 1
  Score at Week 12=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 0 | 0
  Score at Week 12=3 (Severe): Score at Baseline=3 (Severe) | 1 | 1 | 9
  Score at Week 12=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=4 (Very Severe): number analyzed (Participants) | 1 | 1 | 0
  Score at Week 12=4 (Very Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 |
  Score at Week 12=4 (Very Severe): Score at Baseline=1 (Mild) | 0 | 0 |
  Score at Week 12=4 (Very Severe): Score at Baseline=2 (Moderate) | 0 | 0 |
  Score at Week 12=4 (Very Severe): Score at Baseline=3 (Severe) | 0 | 0 |
  Score at Week 12=4 (Very Severe): Score at Baseline=4 (Very Severe) | 1 | 1 |
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.666, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.812, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.834, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.841, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.893, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.907, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

16. Secondary Outcome: Number of Participants by Patient Global Impression-Severity (PGI-S) (Global Severity) Score Categories Relative to Baseline
Description: The participant assessed the severity of their disease overall using the PGI-S 5-point scale where: 0=No symptoms, 1=Mild, 2=Moderate, 3=Severe and 4=Very severe. The number of participants by PGI-S score category is reported relative to their PGI-S score at Baseline. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Score at Week 2=1 (Mild): number analyzed (Participants) | 7 | 4 | 5
  Score at Week 2=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=1 (Mild): Score at Baseline=1 (Mild) | 5 | 1 | 2
  Score at Week 2=1 (Mild): Score at Baseline=2 (Moderate) | 2 | 3 | 3
  Score at Week 2=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 | 0
  Score at Week 2=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=2 (Moderate): number analyzed (Participants) | 16 | 8 | 17
  Score at Week 2=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=2 (Moderate): Score at Baseline=1 (Mild) | 2 | 0 | 0
  Score at Week 2=2 (Moderate): Score at Baseline=2 (Moderate) | 11 | 5 | 16
  Score at Week 2=2 (Moderate): Score at Baseline=3 (Severe) | 3 | 3 | 1
  Score at Week 2=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=3 (Severe): number analyzed (Participants) | 3 | 1 | 4
  Score at Week 2=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 2=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 0
  Score at Week 2=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 0 | 0
  Score at Week 2=3 (Severe): Score at Baseline=3 (Severe) | 3 | 1 | 4
  Score at Week 2=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 2=4 (Very Severe): number analyzed (Participants) | 1 | 0 | 0
  Score at Week 2=4 (Very Severe): Score at Baseline=0 (No Symptoms) | 0 |  |
  Score at Week 2=4 (Very Severe): Score at Baseline=1 (Mild) | 0 |  |
  Score at Week 2=4 (Very Severe): Score at Baseline=2 (Moderate) | 0 |  |
  Score at Week 2=4 (Very Severe): Score at Baseline=3 (Severe) | 1 |  |
  Score at Week 2=4 (Very Severe): Score at Baseline=4 (Very Severe) | 0 |  |
  Score at Week 7=1 (Mild): number analyzed (Participants) | 5 | 3 | 4
  Score at Week 7=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 7=1 (Mild): Score at Baseline=1 (Mild) | 4 | 1 | 2
  Score at Week 7=1 (Mild): Score at Baseline=2 (Moderate) | 1 | 2 | 2
  Score at Week 7=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 | 0
  Score at Week 7=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 7=2 (Moderate): number analyzed (Participants) | 18 | 7 | 16
  Score at Week 7=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 7=2 (Moderate): Score at Baseline=1 (Mild) | 2 | 0 | 0
  Score at Week 7=2 (Moderate): Score at Baseline=2 (Moderate) | 12 | 4 | 14
  Score at Week 7=2 (Moderate): Score at Baseline=3 (Severe) | 4 | 3 | 2
  Score at Week 7=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 7=3 (Severe): number analyzed (Participants) | 3 | 3 | 4
  Score at Week 7=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 7=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 0
  Score at Week 7=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 2 | 1
  Score at Week 7=3 (Severe): Score at Baseline=3 (Severe) | 3 | 1 | 3
  Score at Week 7=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=1 (Mild): number analyzed (Participants) | 6 | 3 | 4
  Score at Week 12=1 (Mild): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=1 (Mild): Score at Baseline=1 (Mild) | 4 | 1 | 2
  Score at Week 12=1 (Mild): Score at Baseline=2 (Moderate) | 2 | 2 | 2
  Score at Week 12=1 (Mild): Score at Baseline=3 (Severe) | 0 | 0 | 0
  Score at Week 12=1 (Mild): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=2 (Moderate): number analyzed (Participants) | 16 | 7 | 18
  Score at Week 12=2 (Moderate): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=2 (Moderate): Score at Baseline=1 (Mild) | 2 | 0 | 0
  Score at Week 12=2 (Moderate): Score at Baseline=2 (Moderate) | 10 | 4 | 15
  Score at Week 12=2 (Moderate): Score at Baseline=3 (Severe) | 4 | 3 | 3
  Score at Week 12=2 (Moderate): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
  Score at Week 12=3 (Severe): number analyzed (Participants) | 2 | 2 | 2
  Score at Week 12=3 (Severe): Score at Baseline=0 (No Symptoms) | 0 | 0 | 0
  Score at Week 12=3 (Severe): Score at Baseline=1 (Mild) | 0 | 0 | 0
  Score at Week 12=3 (Severe): Score at Baseline=2 (Moderate) | 0 | 1 | 0
  Score at Week 12=3 (Severe): Score at Baseline=3 (Severe) | 2 | 1 | 2
  Score at Week 12=3 (Severe): Score at Baseline=4 (Very Severe) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.216, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.215, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.411, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.194, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.408, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

17. Secondary Outcome: Number of Participants by CGI-S (Upper Extremity Functional Severity) Score Categories Relative to Baseline
Description: The clinician used the CGI-S scale to assess the severity of the participant's upper extremity function on a 5-point scale where: 0=Not impaired, 1=Mildly impaired, 2=Moderately impaired, 3=Severely impaired and 4=Very severely impaired. The number of participants by CGI-S score category is reported relative to their CGI-S score at Baseline. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Baseline and Week 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Score at Week 2=1 (Mildly Impaired): number analyzed (Participants) | 13 | 5 | 13
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 13 | 3 | 11
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 2 | 1
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 1
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 2=2 (Moderately Impaired): number analyzed (Participants) | 14 | 7 | 11
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 2 | 2 | 2
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 11 | 5 | 8
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 1 | 0 | 0
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 1
  Score at Week 7=1 (Mildly Impaired): number analyzed (Participants) | 12 | 7 | 9
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 10 | 4 | 9
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 2 | 3 | 0
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 7=2 (Moderately Impaired): number analyzed (Participants) | 14 | 6 | 13
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 4 | 1 | 3
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 9 | 5 | 8
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 1 | 0 | 1
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 1
  Score at Week 12=1 (Mildly Impaired): number analyzed (Participants) | 12 | 5 | 10
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 10 | 3 | 9
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 2 | 2 | 0
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 1
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): number analyzed (Participants) | 12 | 6 | 13
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 4 | 1 | 4
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 7 | 5 | 8
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 1 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.406, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.235, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.225, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.434, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.249, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.380, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

18. Secondary Outcome: Number of Participants by PGI-S (Upper Extremity Functional Severity) Score Categories
Description: The participant assessed the severity of their upper extremity function using the PGI-S 5-point scale where: 0=Not impaired, 1=Mildly impaired, 2=Moderately impaired, 3=Severely impaired and 4=Very severely impaired. The number of participants by PGI-S score category is reported relative to their PGI-S score at Baseline. Only those score categories reported for at least one participant at the given time-point are presented.
Time Frame: Baseline and Weeks 2, 7, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  Score at Week 2=0 (Not Impaired): number analyzed (Participants) | 0 | 1 | 0
  Score at Week 2=0 (Not Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 2=0 (Not Impaired): Score at Baseline=1 (Mildly Impaired) | 0 | 1 | 0
  Score at Week 2=0 (Not Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 0 | 0
  Score at Week 2=0 (Not Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 2=0 (Not Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 2=1 (Mildly Impaired): number analyzed (Participants) | 14 | 4 | 14
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 1 | 1 | 0
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 11 | 2 | 9
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 2 | 1 | 2
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 3
  Score at Week 2=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 2=2 (Moderately Impaired): number analyzed (Participants) | 12 | 6 | 12
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 1 | 1 | 5
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 11 | 5 | 6
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 1
  Score at Week 2=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 2=3 (Severely Impaired): number analyzed (Participants) | 0 | 1 | 0
  Score at Week 2=3 (Severely Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 2=3 (Severely Impaired): Score at Baseline=1 (Mildly Impaired) | 0 | 0 | 0
  Score at Week 2=3 (Severely Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 1 | 0
  Score at Week 2=3 (Severely Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 2=3 (Severely Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 7=0 (Not Impaired): number analyzed (Participants) | 1 | 0 | 1
  Score at Week 7=0 (Not Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 7=0 (Not Impaired): Score at Baseline=1 (Mildly Impaired) | 1 | 0 | 0
  Score at Week 7=0 (Not Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 0 | 0
  Score at Week 7=0 (Not Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 1
  Score at Week 7=0 (Not Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 7=1 (Mildly Impaired): number analyzed (Participants) | 11 | 5 | 16
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 1 | 1 | 0
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 8 | 1 | 9
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 2 | 3 | 5
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 2
  Score at Week 7=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 7=2 (Moderately Impaired): number analyzed (Participants) | 14 | 7 | 7
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 3 | 3 | 4
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 11 | 4 | 3
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 7=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 7=3 (Severely Impaired): number analyzed (Participants) | 0 | 1 | 0
  Score at Week 7=3 (Severely Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 7=3 (Severely Impaired): Score at Baseline=1 (Mildly Impaired) | 0 | 0 | 0
  Score at Week 7=3 (Severely Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 1 | 0
  Score at Week 7=3 (Severely Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 7=3 (Severely Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 12=0 (Not Impaired): number analyzed (Participants) | 1 | 0 | 0
  Score at Week 12=0 (Not Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 12=0 (Not Impaired): Score at Baseline=1 (Mildly Impaired) | 1 | 0 | 0
  Score at Week 12=0 (Not Impaired): Score at Baseline=2 (Moderately Impaired) | 0 | 0 | 0
  Score at Week 12=0 (Not Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 12=0 (Not Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 12=1 (Mildly Impaired): number analyzed (Participants) | 13 | 3 | 16
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=0 (Not Impaired) | 1 | 0 | 0
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=1 (Mildly Impaired) | 9 | 2 | 11
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=2 (Moderately Impaired) | 3 | 1 | 2
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 3
  Score at Week 12=1 (Mildly Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): number analyzed (Participants) | 10 | 9 | 8
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=0 (Not Impaired) | 0 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=1 (Mildly Impaired) | 2 | 2 | 2
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=2 (Moderately Impaired) | 8 | 7 | 6
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=3 (Severely Impaired) | 0 | 0 | 0
  Score at Week 12=2 (Moderately Impaired): Score at Baseline=4 (Very Severely Impaired) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Week 2; Test type: Superiority; p = 0.422, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Week 2; Test type: Superiority; p = 0.226, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Week 7; Test type: Superiority; p = 0.639, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Week 7; Test type: Superiority; p = 0.094, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Week 12; Test type: Superiority; p = 0.516, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Week 12; Test type: Superiority; p = 0.266, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]

19. Secondary Outcome: Change From Baseline in the ADL Component Score for Upper Limb Function Items of the FARS
Description: The ADL component of the FARS includes 9 subscales: speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function. Items 3 to 5 are directly related to upper limb function. Each of these subscales is rated on a 5-point scale where 0=normal to 4=severe disability/inability to carry out activity independently for a total possible score of 0 to 12, with higher scores representing greater disability/dependency. A negative change from Baseline indicates improvement. Change from Baseline in Friedreich ataxia rating scale activities of daily living (FARS ADL) upper limb function items was analyzed using MMRM ANCOVA with Baseline FARS ADL as a covariate; pooled site, visit, treatment, and ambulation status (randomization factor) as fixed factors; and treatment-by-visit and Baseline FARS ADL-by-visit interactions.
Time Frame: Baseline and Weeks 2, 7 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 27 | 13 | 26
  Change from Baseline at Week 2 | -0.21 (0.213) | -0.40 (0.308) | 0.34 (0.212)
  Change from Baseline at Week 7: number analyzed (Participants) | 26 | 13 | 24
  Change from Baseline at Week 7 | -0.17 (0.202) | -0.14 (0.289) | 0.16 (0.203)
  Change from Baseline at Week 12: number analyzed (Participants) | 24 | 12 | 24
  Change from Baseline at Week 12 | -0.15 (0.240) | -0.05 (0.345) | 0.19 (0.240)
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.299, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.19, 90% CI 2-sided [-0.80 to 0.41], Standard Error of Mean 0.362
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 2; Test type: Superiority; p = 0.967, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.55, 90% CI 2-sided [0.06 to 1.04], Standard Error of Mean 0.293
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.529, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.02, 90% CI 2-sided [-0.54 to 0.59], Standard Error of Mean 0.338
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 7; Test type: Superiority; p = 0.880, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.33, 90% CI 2-sided [-0.13 to 0.80], Standard Error of Mean 0.279
Statistical Analysis 5: Comparison: Placebo vs TAK-831 75 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.599, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.10, 90% CI 2-sided [-0.58 to 0.79], Standard Error of Mean 0.408
Statistical Analysis 6: Comparison: Placebo vs TAK-831 300 mg; Change from Baseline at Week 12; Test type: Superiority; p = 0.846, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.34, 90% CI 2-sided [-0.21 to 0.90], Standard Error of Mean 0.333

20. Secondary Outcome: Number of Participants With at Least a 15 Percent (%) or at Least a 20% Reduction in 9-HPT Completion Time From Baseline
Description: The 9-HPT-1 is a measure of timed upper extremity (arm and hand) function and manual dexterity. The participant picks up pegs 1 at a time (9 in total), using 1 hand only, and places them into holes on the board as quickly as possible, in any order until all holes are filled. Then, without pausing, the participant removes the pegs 1 at a time and returns them as quickly as possible. Each participant performs this task twice with each hand separately. Results on both tests are then averaged for an overall task completion time.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
Number analyzed (Participants) | 27 | 14 | 26
Participants
  At Least 15% Reduction from Baseline | 3 | 0 | 0
  At Least 20% Reduction from Baseline | 2 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs TAK-831 75 mg; At Least 15% Reduction from Baseline; Test type: Superiority; p > 0.999, Fisher Exact — P-value was from Fisher's exact test. Odds ratio was obtained from Cochran-Mantel-Haenszel with ambulation status at randomization as a stratification factor; Odds Ratio (OR) = 0.00
Statistical Analysis 2: Comparison: Placebo vs TAK-831 300 mg; At Least 15% Reduction from Baseline; Test type: Superiority; p > 0.999, Fisher Exact — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 0.00
Statistical Analysis 3: Comparison: Placebo vs TAK-831 75 mg; At Least 20% Reduction from Baseline; Test type: Superiority; p > 0.999, Fisher Exact — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 0.00
Statistical Analysis 4: Comparison: Placebo vs TAK-831 300 mg; At Least 20% Reduction from Baseline; Test type: Superiority; p > 0.999, Fisher Exact — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 0.00

ADVERSE EVENTS:
Time Frame: First dose of study drug to up to 17 days past last dose (up to 14.4 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
  Safety analysis set included all randomized participants who received at least 1 dose of double-blind study medication.
Arm/Group | Placebo | TAK-831 75 mg | TAK-831 300 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/14 | 0/26
Other Adverse Events (participants affected / at risk) | 21/27 | 10/14 | 24/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | TAK-831 75 mg (N=14) | TAK-831 300 mg (N=26)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Altered visual depth perception (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 8
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Fatigue (General disorders) | 4 | 0 | 3
Pain (General disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 1 | 6
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 4 | 11
Dizziness (Nervous system disorders) | 2 | 1 | 1
Aphonia (Nervous system disorders) | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 2
Coordination abnormal (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03214588/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03214588/SAP_001.pdf